CLINICAL TRIAL: NCT02555293
Title: Administration of Rifaximin to Improve Liver Regeneration and Outcome Following Major Liver Resection
Acronym: ARROW
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Prematurely terminated due to organisational reasons
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTC-A 13-129
Record Dates: First submitted 2015-09-14; First posted 2015-09-21 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2020-10

CONDITIONS: Malignant Liver Disease; Major Liver Resection
Keywords: Liver resection; fibrosis; inflammation; Rifaximin
MeSH Terms: conditions — Fibrosis; Inflammation | interventions — Rifaximin

ARMS (2):
- film-coated Rifaximin (550 mg) (Experimental): (550 mg) tablet twice daily for at least 14 days but up to 28 days dependent on the need for a PVE and the period between PVE (portal vein embolization) or randomization and surgery. Preoperative Rifaximin treatment in case of a PVE will start the day after PVE and will last for 14-21 days. In case patients are not pre-treated with a PVE they will receive Rifaximin for 7-10 days prior to surgery. Regardless of PVE, patients will receive additional Rifaximin treatment the first 7 days postoperatively.
  Interventions: Drug: XIFAXAN® (Rifaximin)
- standard therapy (No Intervention): Patients directed to the control group will not receive Rifaximin.

INTERVENTIONS:
Drug: XIFAXAN® (Rifaximin)
  Other Names: NDA 22-554
  Arms: film-coated Rifaximin (550 mg)

SUMMARY:
Surgery is in almost all cases the only potentially curative treatment option for patients with primary or secondary malignancies of the liver. However, in most cases oncological resections ("R0-resections") can only be achieved by performing major liver resections (4 or more liver segments), which is related to considerable postoperative complications such as systemic infections and postoperative liver insufficiency (postresectional liver failure (PRLF)). Despite optimized preoperative and postoperative strategies of care presently, up to 32-55% of patients display severs postoperative complications (Clavien score ≥ 3a) and 5% even suffer from a severe PRLF. Recent observations in murine disease models as well as human patients suggested that postoperative alterations of hemodynamics within the portal vein tract as well as postoperative modulations of the immune response facilitates the translocation of gut bacteria in the blood, leading to systemic infections and sepsis. Moreover it became apparent that inflammatory mediators, released by the gut microbiota might negatively affect postoperative liver regeneration. Rifaximin (Xifaxan®) is a novel and potent, semisynthetic antibiotic that efficiently acts against most enteric bacteria and significantly reduced liver inflammation and liver fibrosis in animal studies. Moreover, Rifaximin is very well tolerated, even in patients with liver insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing a liver resection of at least 4 segments
2. Age > 18 years < 80 years
3. BMI 18-40
4. Patients with ASA (American Society of Anesthesiologists) I-III
5. Written informed consent prior to study participation

Exclusion Criteria:

1. Patients with ASA IV-V
2. Contraindication for MRI (see 5.4.3)
3. Underlying chronic liver disease such as severe fibrosis or liver cirrhosis
4. Need for procedures additive to partial liver resection
5. Participation in other liver related trials
6. BMI > 40
7. Previous liver transplantation or porto-systemic shunt
8. Concomitant acute infectious diseases
9. Renal insufficiency
10. Hypersensitivity to Rifaximin
11. Concomitant HIPEC (hypertherme intraperitoneale chemoperfusion) treatment
12. ALPPS (associating liver partition and portal vein ligation for staged hepatectomy)
13. Pregnant females as determined by positive [serum or urine] hCG (human chorionic gonadotropin) test at Screening or prior to dosing. Participants of child-bearing age should use adequate contraception as defined in the study protocol.
14. Lactating females
15. The subject has a history of any other illness, which, in the opinion of the investigator, might pose an unacceptable risk by administering study medication.
16. The subject received an investigational drug within 30 days prior to inclusion into this study
17. The subject has any current or past medical condition and/or required medication to treat a condition that could affect the evaluation of the study
18. The subject is unwilling or unable to follow the procedures outlined in the protocol
19. The subject is mentally or legally incapacitated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2016-02; Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Effect of Rifaximin on postoperative liver function | Postoperative day 7 in relation to postoperative day 4
  LiMAx liver function percentage increase on postoperative day 7 in relation to LiMAx value on postoperative day 4 compared to a control group without Rifaximin treatment.
  LiMAx will be made after at least 14 days but up to 28 days of treatment (control group analogue) dependent on the need for a PVE and the period between PVE or randomization and surgery

SECONDARY OUTCOMES:
postoperative morbidity/Complications | minimum 14 days after liver resection
  Complications will be scored using the Clavien-Dindo scoring system and a liver-specific-composite-endpoint for the duration of hospital stay, an expected average of minimum 14 days
Liver volume percentage increase | 14 up to 21 days before liver resection at baseline and 7 days after the operation
  MRI volumetry:
  pre- and postoperative comperative measurements mainly based on suitable, preoperatively and routinely done MRI/CT-images. On postoperative day 7 as tudy related MRI will be done if no CT/MRI images available routinely done 1 day before or one day after visit 5
liver function percentage increase | 14 up to 21 days before liver resection at baseline (all), on preoperative day 1 (PVE group only) and on postoperative day 4 and day 7 (all)
  LiMAx-test:
  LiMAx liver function testing will be performed before surgery and on postoperative days 4 and 7 to evaluate functional recovery after liver resection.
Time to functional recovery | minimum 14 days starting on operation day
  The evaluation of time to functional recovery will start on POD 0 and will be scored daily until discharge from the hospital with the following criteria
  * Adequate pain control on oral analgesics only
  * Eating and drinking properly without the need of IV fluids
  * Independently mobile or mobile at preoperative level
  * Standard laboratory tests and liver function returning to normal level When all of these criteria are met, we consider a patient functional recovered.

CONTACTS AND LOCATIONS:
Locations (1):
- RWTH Aachen University, Aachen, Germany

REFERENCES:
- [Derived] Bednarsch J, Czigany Z, Loosen SH, Heij L, Ruckgaber L, Maes H, Krause JP, Reen M, Toteva B, Vosdellen T, Bruners P, Lang SA, Ulmer TF, Roderburg C, Luedde T, Neumann UP. Perioperative rifaximin is not associated with enhanced functional and volumetric recovery after major liver resection. Sci Rep. 2021 Sep 9;11(1):17936. doi: 10.1038/s41598-021-97442-w. PMID 34504196